CLINICAL TRIAL: NCT06315621
Title: Deviation Parameters of Intraoral Scanning with and Without Artificial Markers Versus Conventional Impression of Total, Partial and Congenital Nasal Defects: a Pilot Non-Randomized Clinical Trial
Brief Title: Deviation Parameters of Intraorfal Scanning in Capturing Different Intraoral Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatima Elmougi, Doctor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 36124
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Nasal Defect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical impression (Active Comparator)
  Interventions: Device: Physical Impression
- Scanning using intraoral scanner without markers (Experimental)
  Interventions: Device: Scanning using intraoral scanner without markers
- Scanning using Intraoral scanner with markers (Experimental)
  Interventions: Device: Scanning using intraoral scanner with markers

INTERVENTIONS:
Device: Scanning using intraoral scanner with markers — Scanning different types of nasal defects using intraoral scanner with skin markers.
  Arms: Scanning using Intraoral scanner with markers
Device: Scanning using intraoral scanner without markers — Scanning different types of nasal defects using intraoral scanner without skin markers.
  Arms: Scanning using intraoral scanner without markers
Device: Physical Impression — Recording different types of nasal defects using physical impressions
  Arms: Physical impression

SUMMARY:
For all participants, a conventional facial impression will be done using silicone material then poured and scanned using a desktop scanner which represented the control group (Group 1).

Group 2, involves nasal defects which will be optically scanned using IOS(medit 700 wireless) without facial markers Group 3 involves nasal defects which will be optically scanned using IOS(medit 700 wireless) with facial markers.

STL files of the facial scans and scanned cast obtained from the impression will be exported and saved to be used later for outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* isolated nasal defects either, total or subtotal.
* congenitally missing external nose with healthy and intact remaining facial structures.

Exclusion Criteria:

* Any debilitating medical condition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Dimensional accuracy of intraoral scanners | Day 0
  measuring dimensional accuracy of diffrent scanning techniques using intraoral scanners

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No